CLINICAL TRIAL: NCT04459546
Title: The Effect of Rational Drug Use and Symptom Control Training on Self-efficacy, Emotional Status and Clinical Parameters in COPD (Chronic Obstructive Pulmonary Disease)
Brief Title: Nurse-led COPD Self-management Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Şenay Takmak, PhD student, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 60116787-020/4317
Record Dates: First submitted 2020-06-24; First posted 2020-07-07 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: COPD; COPD Exacerbation
Keywords: COPD; nursing; self-efficacy; self-management
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: Randomized controlled pre-post test design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Study group intervention consists patient education, training booklet and 3 month follow-up.
  Interventions: Behavioral: patient education, training booklet, 3 months tele health
- Control group (No Intervention): Control group received only general care

INTERVENTIONS:
Behavioral: patient education, training booklet, 3 months tele health — Patient education includes general disease information, COPD self-management and symptom control. The education face-to-face and practical training was provided by the researcher. The training booklet was prepared by the researcher. The readability of the booklet was very easy and its comprehensibility was tested by pre-application. Tele monitoring was done by the researcher for support and motivation. The participants were called 4 times by phone.
  Arms: Study group

SUMMARY:
Introduction: Chronic Obstructive Pulmonary Disease (COPD) disease highest mortality and morbidity of respiratory diseases that third cause of death in the world and Turkey.

Purpose: Purpose of study improve self-efficacy, anxiety/depression, symptom control and exercise capacity, reduce use of health care of COPD patients.

Method: The study was conducted with a randomized controlled design. This study were included 41 COPD patients (İntervention=20, Control=21). Data collection tools were patient description form, COPD Self-Efficacy Scale (CSES), COPD Assessment Test (CAT), Hospital Anxiety Depression Scale (HAD), 6-Minute Walk Test (MWT) and tele-health form. Intervention consists patient education, training booklet and 3 month follow-up. Control group patients received only general care. The final test was performed three months later.

DETAILED DESCRIPTION:
The skills and the knowledge necessary in COPD management and interventions required to develop this skill have conceptualized as self-management. The complex structure of COPD self-management includes medication compliance, smoking cessation, maintaining and increasing exercise capacity, regulating nutrition, healthy lifestyle changes, vaccination and symptom management.

According to the GOLD (2017) report, copd self-management cannot be achieved only with didactic teaching. Skill acquisition, behavior change and motivational interventions should be applied with education. Among these interventions, action plans are among the tools frequently used in preventing tele-health COPD attacks. Action plans can be used effectively in COPD to prevent attacks, symptom management and reduce the risk of anxiety / depression. One objectives of self-management is to reduce use of health care. Symptom management; It has been stated that it is effective in reducing hospitalization and days of hospitalization especially in patients with COPD diseases.

In studies involving self-management in COPD, self-management interventions increase health-related quality of life, control symptom, reduce the risk of anxiety / depression, increase self-efficacy, reduce respiratory hospital stays, reduce severity and duration of attacks, and reduce mortality at low impact. It is stated that the interventions made in the GOLD (2017) report provide improvements for health-related quality of life and patient outcomes. Because of self-management is a multi-component concept, variety in type of intervention and follow-up make it difficult to reach generalizable evidence.

Although many health professionals work with patients with COPD, self-management interventions are known to be carried out mostly by nurses or by multidisciplinary groups involving nurses.

This study is an example of applicable self-management intervention in terms of disease information and general management, rational drug use, symptom control training and evaluation with medium-term monitoring. It can contribute to literature in terms of determining the effect of nurse-managed self-management intervention.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of COPD
* Being inpatient at chest diseases clinic
* Being literate
* Able to use a telephone
* No communication disabilities
* Being volunteers

Exclusion Criteria:

* Having mental illness
* Respiratory comorbidity (lung cancer, interstitial lung disease, pulmonary tuberculosis),
* Unable to attend the post-tests
* Not reachable by phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-02-17 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
COPD Self-Efficacy Score | Change from baseline COPD self-efficacy score at 3 months
  Scales were filled in by interviewing each participant.Scoring is done between 1-5 points. Increased score indicates an increase in self-efficacy in coping with respiratory distress.
COPD Assessment Test Score | Change from baseline COPD assessment test score at 3 months
  Scales were filled in by interviewing each participant.Scoring is done between 0-40 points. Increased points indicate that the severity of the disease decreases.
Anxiety Depression Score | Change from baseline anxiety depression test score at 3 months
  Scales were filled in by interviewing each participant. Turkey cut-off score of the scale used for anxiety, 10, were found to be 7 for depression. Participants who scored above these points were evaluated as risky.
6-Minute Walk Test | Change from baseline 6-minute walk distance at 3 months
  Each participant received a 6-minute walk test as recommended by the AmericanThoracic Society.

SECONDARY OUTCOMES:
Number of health care uses | Change in the number of initial health care use in the 3rd month
  According to the patient's declaration, emergency room visit, chest diseases outpatient clinic and hospitalizations associated with respiration

CONTACTS AND LOCATIONS:
Overall Officials: Nevin K Kurban, Prof. Dr., Study Director — Consultant, Responsible researcher; Şenay Takmak, pHd, Principal Investigator — pHd student, Assistant researcher
Locations (1):
- Denizli Public Hospitals Association, Buldan Chest Diseases Hospital, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study results will be announced in a publication.
Supporting Information: Study Protocol, SAP
Time Frame: Findings can be shared after the study has been published.
Access Criteria: The sociodemographic and disease-related characteristics of the participants, the pre-post-test findings including the answers to the research questions and statistical analyzes will be shared.
URL: http://acikerisim.pau.edu.tr/xmlui/handle/11499/28554

REFERENCES:
- [Background] Kasikci MK. Using self-efficacy theory to educate a patient with chronic obstructive pulmonary disease: A case study of 1-year follow-up. Int J Nurs Pract. 2011 Feb;17(1):1-8. doi: 10.1111/j.1440-172X.2010.01898.x. PMID 21251148
- [Background] Global Initiative for Chronic Obstructive Lung Disease, From the Global Strategy for the Diagnosis, Management and Prevention of COPD, GOLD 2017, p.139. https://goldcopd.org/wp-content/uploads/2017/02/wms-GOLD-2017-FINAL.pdf (access date: 10.08.2018)
- [Background] Harrison SL, Janaudis-Ferreira T, Brooks D, Desveaux L, Goldstein RS. Self-management following an acute exacerbation of COPD: a systematic review. Chest. 2015 Mar;147(3):646-661. doi: 10.1378/chest.14-1658. PMID 25340578
- [Result] Trappenburg JC, Koevoets L, de Weert-van Oene GH, Monninkhof EM, Bourbeau J, Troosters T, Verheij TJ, Lammers JW, Schrijvers AJ. Action Plan to enhance self-management and early detection of exacerbations in COPD patients; a multicenter RCT. BMC Pulm Med. 2009 Dec 29;9:52. doi: 10.1186/1471-2466-9-52. PMID 20040088